CLINICAL TRIAL: NCT00003173
Title: High-Dose Thiotepa With Autologous Stem Cell Rescue in Patients With Malignancies Refractory to Conventional Chemotherapy
Brief Title: High-Dose Thiotepa Plus Peripheral Stem Cell Transplantation in Treating Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-089; P30CA008748 (NIH); MSKCC-97089A3; NYU-97-7; NCI-G97-1366
Record Dates: First submitted 1999-11-01; First posted 2003-04-23 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Ovarian Cancer; Retinoblastoma; Testicular Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: intraocular retinoblastoma; recurrent retinoblastoma; childhood central nervous system germ cell tumor; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; childhood germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; extragonadal germ cell tumor; adult central nervous system germ cell tumor; childhood teratoma; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Ovarian Neoplasms; Retinoblastoma; Testicular Germ Cell Tumor; Testicular Neoplasms; Teratoma; Ovarian Germ Cell Cancer | interventions — Filgrastim; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: thiotepa
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose thiotepa plus peripheral stem cell transplantation in treating patients with refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy and toxicity of sequential cycles of high dose thiotepa with stem cell rescue and filgrastim in patients with malignancies refractory to conventional chemotherapy or for whom conventional therapy is not available.
* Evaluate the effectiveness of autologous stem cells in restoring hematopoiesis following high dose thiotepa.

OUTLINE: Patients are stratified by type of tumor (neuroectodermal CNS tumor vs non-neuroectodermal CNS tumor vs non-CNS small round blue cell tumor vs other non-CNS tumor).

Autologous stem cells are obtained prior to the administration of thiotepa. Patients who do not have peripheral blood stem cells available may undergo a bone marrow harvest instead. Thiotepa is administered as a 3 hour infusion daily for 3 consecutive days. Stem cells are reinfused approximately 72 hours following the completion of thiotepa. Filgrastim is administered the day following reinfusion of stem cells and continues until there is sufficient hematopoietic recovery.

The second course of thiotepa is administered 4 weeks following the first course in patients who have responding or stable disease, adequate stem cells, and no unacceptable toxicity. Patients receive a maximum of 2 courses.

PROJECTED ACCRUAL: Approximately 36 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Malignant solid tumors
* Must have failed conventional treatment or for whom conventional therapy is not available
* Measurable disease by MRI or CT scan

  * Intraocular retinoblastomas may be measured by direct visualization
  * Germ cell tumors may be measured by tumor markers
* No known bone marrow involvement

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Lansky 60-100% for patients 16 and under
* Karnofsky 60-100% for patients over 16

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3
* If parameters not met, must have adequate stem cell yield

Hepatic:

* Bilirubin no greater than 1.5 times the upper limit of normal (ULN)
* SGOT and SGPT no greater than 2.5 times the ULN (unless liver involvement by tumor)

Renal:

* Creatinine within normal limits OR
* Creatinine clearance at least 70 mL/min

Cardiovascular:

* Fractional shortening greater than 28% on echocardiogram OR
* Ejection fraction at least 55% on RNCA prior to first cycle of thiotepa

Pulmonary:

* DLCO greater than 55% of predicted (only required if there is clinical evidence of pulmonary dysfunction)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior bone marrow or peripheral blood stem cell rescue allowed

Chemotherapy:

* At least 4 weeks since prior chemotherapy if absolute neutrophil count is less than 1,000/mm^3 or platelet count is less than 75,000/mm^3, and recovered (i.e. adequate stem cells collected to predict hematopoietic recovery)
* No concurrent chemotherapy except for dexamethasone for antiedema effects

Endocrine therapy:

* No concurrent use of corticosteroids used solely as antiemetics

Radiotherapy:

* At least 4 weeks since radiotherapy if absolute neutrophil count is less than 1,000/mm^3 or platelet count is less than 75,000/mm^3, and recovered (i.e. adequate stem cells collected to predict hematopoietic recovery)
* No concurrent radiotherapy

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1997-09; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York